CLINICAL TRIAL: NCT03190395
Title: Compared With 2 Different Ablation Strategies Clinical Outcome for Treating Patients With Paroxysmal Atrial Fibrillation，Prospective Randomised Study
Brief Title: Compared With 2 Different Ablation Strategies Clinical Outcome for Treating Patients With Paroxysmal Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1033415
Record Dates: First submitted 2017-06-13; First posted 2017-06-16 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-03

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Paroxysmal Atrial Fibrillation; Circumferential Pulmonary Vein Isolation(CPVI); Leftatrium Roofline Ablation(LARA); Longterm success rate
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Contorol Group:Pure Circumferential pulmonary vein isolation(CPVI) Experimental Group:Circumferential pulmonary vein isolation combine with Left atrium roofline ablation(CPVI+LARA)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPVI Group (Experimental): CPVI Group: Pure Circumferential pulmonary vein isolation(CPVI)
  Interventions: Procedure: CPVI Group
- CPVI+LARA Group (Active Comparator): CPVI+LARA Group: Circumferential pulmonary vein isolation combine with Left Atrium Roofline Ablation
  Interventions: Procedure: CPVI+LARA Group

INTERVENTIONS:
Procedure: CPVI Group — CPVI Group:The ablation strategy of Circumferential pulmonary vein isolation (CPVI)will be operated on 60 patients with paroxysmal atrial fibrillation.
  Other Names: Pure Circumferential pulmonary vein isolation
  Arms: CPVI Group
Procedure: CPVI+LARA Group — CPVI+LARA Group: The ablation strategy of Circumferential pulmonary vein isolation combine with Left atrium roofline ablation(CPVI+LARA) will be operated on 60 patients with paroxysmal atrial fibrillation.
  Other Names: Circumferential pulmonary vein isolation combine with Left atrium roofline ablation
  Arms: CPVI+LARA Group

SUMMARY:
Atrial fibrillation (AF) is the most serious atrial electrical activity disorders, is also one of the common tachyarrhythmias.Circumferential pulmonary Vein Isolation (CPVI) is considered to be the cornerstone of paroxysmal atrial fibrillation ablation, but recently reported in the literature that pure CPVI treatment for paroxysmal atrial fibrillation the 5-year success rate as low as 46.6%, and the incidence of atrial reentry tachycardia is also high in the follow-up period. Therefore it is necessary for us to explore whether the success rate of CPVI combined with Leftatrium Roofline Ablation (CPVI + LARA) for paroxysmal atrial fibrillation is higher than the pure CPVI.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) refers to the orderly loss of atrial electrical activity, replaced by rapid and disorderly atrial fibrillation wave, is the most acute atrial electrical activity disorders, is also one of the common tachyarrhythmias. So far, the mechanism of atrial fibrillation has not yet been completely clarified. At present, there are various mechanisms to participate in the occurrence and maintenance of atrial fibrillation, which mainly involves two aspects. One is the triggering factor of atrial fibrillation, and the other is the occurrence and maintenance of atrial fibrillation (substrate). Trigger factors are varied, including sympathetic and parasympathetic stimulation, bradycardia, atrial premature beats or tachycardia, atrioventricular bypass and acute atrial pull, etc, which pulmonary vein electrical activity triggered the most common, but also is an most important theoretical Basis for the Radiofrequency Catheter Ablation of Atrial Fibrillation . Substrate is a necessary condition for the onset and maintenance of atrial fibrillation. Electrical remodeling and structural remodeling are by shortening the atrial effective refractory period. Atrial dilatation and atrial fibrosis play a major role in the formation of atrial fibrillation reentry.Circumferential pulmonary Vein Isolation (CPVI) is considered to be the cornerstone of paroxysmal atrial fibrillation ablation, but recently reported in the literature that pure CPVI treatment for paroxysmal atrial fibrillation the 5-year success rate as low as 46.6%, and the incidence of atrial reentry tachycardia is also high in the follow-up period. Therefore it is necessary for us to explore whether the success rate of CPVI combined with Leftatrium Roofline Ablation (CPVI + LARA) for paroxysmal atrial fibrillation is higher than the pure CPVI.

ELIGIBILITY:
Inclusion Criteria:

- (1)Patients between 18-80 year-old with paroxysmal atrial fibrillation have radio frequency ablation operation indication and are willing to require AF ablation therapy.

(2)Voluntary consent of informed consent (3)No AF Ablation history before admission

Exclusion Criteria:

* (1) Permanent or persistent AF (2) The diameter of left atrium >50mm (3) Previous AF/AFL/AT Radio Frequency Ablation (4) Congenital heart disease and/or Cardiac Surgical procedures (5) AF with rheumatic valvular disease (6) LV ejection fraction <45% (7) Intracardiac thrombi

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-20 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Maintenance time of sinus rhythm | The two groups will be assessed from 3 months later operation until the recurrence of atrial fibrillation or up to 36 months after operation
  To evaluate the effectiveness of the ablation operation, we will observe how long will these patients keep sinus rhythm after operation.

SECONDARY OUTCOMES:
The size of the left atrium | Patients's size of the left atrium will be assessed from 3 months later operation until the recurrence of atrial fibrillation or up to 36 months after operation
  The size of the left atrium measured by Transthoracic echocardiography
The Left Ventricular Ejection Fraction | Patients's LV ejection fraction will be assessed from 3 months later operation until the recurrence of atrial fibrillation or up to 36 months after operation
  The Left Ventricular Ejection Fraction measured by Transthoracic echocardiography maybe improve when heart rhytum becom sinus rhytum after ablation operation.

CONTACTS AND LOCATIONS:
Overall Officials: Pingzhen Yang, Doctor, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital,Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No